CLINICAL TRIAL: NCT06784154
Title: The Association of Ectopic Fat and Cardiovascular Disease in People Living With HIV and General Populations: A Cross Sectional Analysis
Brief Title: The Role of Ectopic Fat and Heart Attack Risk in HIV
Acronym: BHIVA
Status: Recruiting | Type: Observational
Sponsor: University of Liverpool (Other)
Responsible Party: Sponsor
Other Study IDs: UOL001832
Record Dates: First submitted 2024-01-30; First posted 2025-01-20 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2024-08

CONDITIONS: Cardiometabolic Syndrome; Hiv
MeSH Terms: conditions — Metabolic Syndrome; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will be taking whole blood for future research purposes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- People living with HIV
  Interventions: Other: Non-interventional
- General population

INTERVENTIONS:
Other: Non-interventional — Non-interventional
  Groups: People living with HIV

SUMMARY:
This study is designed to investigate differences between people living with HIV (PLWHIV) and general populations on how the body utilises and stores energy. This study uses magnetic resonance imaging (MRI) to measure fat around the body organs including the heart and liver. The fat around body organs, also known as visceral fat, is known to be associated with metabolic syndrome and a risk factor for developing heart attacks and strokes.

MRI scans are used frequently in hospitals to diagnose a range of conditions. These scans use radio waves to measure protons in body tissues. The machines can reconstruct tissues using complex algorithms to form composite images of body structures. MRI scans do not use ionising radiation and there is no risk to undertaking an MRI in terms of radiation.

We often use MRI scans to assess the hearts' structure and function. In addition, we can use specific MRI sequences to assess the integrity of heart muscle. Heart MRI is often considered the gold standard imaging technique to assess the heart and heart muscle disease. This sub-study will use multiple MRI sequences to assess the heart and the liver. We are aiming to investigate any changes in heart and liver fat. In addition, we will assess any changes in fat levels within the heart muscle cells whilst also assessing for any change in the way the heart is functioning.

PLWHIV have roughly double the risk of heart attacks compared to general populations. Previous studies have demonstrated that this increased risk may arise from the way in which fat is stored and metabolised in the body. We hope this study will give insight into why HIV-positive individuals have increased risks of heart attacks and how reducing visceral fat may reduce risk. It may lead to further medicines or treatment strategies to reduce the risk of heart attacks in HIV-positive individuals.

DETAILED DESCRIPTION:
PLWHIV have an increased risk of developing cardiovascular disease compared to risk matched HIV-negative patients. CVD is a leading cause of morbidity and mortality in PLWHIV and increasing burden on healthcare systems. One model has suggested that the median age of PLWHIV will increase from 43.9 years in 2010 to 56.6 years in 2030 with 78% being diagnosed with CVD. Traditional risk predication tools have been demonstrated to perform poorly in this patient cohort.

This increased risk may be driven by several factors. Viral related mechanisms, ART, and increased prevalence of traditional risk factors (smoking, poor diet, sedentary lifestyle) act in a synergistic fashion to enhance the cardiovascular risk seen in HIV-positive patients. Recent data has focused on the role of energy metabolism as a mechanistic driver for this excess risk. Accessory proteins from the virus and certain antiretroviral agents are known to induce adipocyte dysfunction through reduction of pre-adipocyte differentiation, muted insulin-sensitivity, increased lipolysis, and mitochondrial stress. The net effect of these changes promotes 'central' storage of energy (fatty acids) in VAT and ectopic fat, of which the principal sites are the hepatic parenchyma (NAFLD) and EAT.

Both NAFLD and EAT are increasingly recognised as risk factors for CVD in both PLWHIV and HIV-negative groups. PLWHIV are 25% more likely to develop NAFLD at normal body weights compared to HIV-negative groups. Our work, and others, have demonstrated a significant association of NAFLD in PLWHIV but less so in HIV-negative groups . EAT volume has again been demonstrated to be associated with CVD in general populations. EAT shares a common microcirculation with the epicardial coronary arteries and exerts influence on vascular function through adipokine secretion, buffering of fatty acids, and secretion of inflammatory cytokines. The close anatomical relationship between EAT and the epicardial coronary arteries may indicate a novel substrate for atherogenesis in the context of EAT dysfunction. Again, our work has demonstrated a strongly significant association between EAT volume and incident CVD.

Emerging imaging studies are utilising cardiac MRS to measure intramyocardial metabolites and associations with health and disease. Cardiac MRS provides the ability to co-localise cardiac anatomy, tissue composition and energetic performance in vivo giving the ability to study the pathophysiology and cell biology of metabolic syndrome, glucose metabolism and ectopic fat deposition. Phosphorus MRS allows quantification of calculation of phosphocreatine to ATP ratio (PCr/ATP) which is a marker of myocardial energetic state. Using phosphorus MR spectroscopy myocardial energetic substrate compromise has been found in diabetic cardiomyopathy. It has also been used to study the effects of SGLT2 inhibitors on cardiac energy substrate utilisation. Proton MR spectroscopy allows quantification of intracellular triglyceride which allows further assessment of the metabolic status of cardiac tissue. Previous work has demonstrated increased cardiac steatosis, on cardiac MR spectroscopy, in HIV-positive patients compared to HIV-negative patients . HIV-positive women increased cardiac steatosis was associated with evidence of cardiac diastolic dysfunction. The use of MRS (proton and 31-P) to study the impact of therapeutic interventions on ectopic fat has never been studied in HIV.

Cardiovascular CT is an important imaging modality with widespread clinical and research utility. It has the ability to inform on multiple metrics of CVD including total plaque volume, non-calcified plaque volume, calcium score (Agatston score), plaque morphology and stenosis grading. The use of these measures as surrogates for CVD risk has been used extensively over the last two decades. This imaging modality is of critical importance to HIV / CVD research as trials powered for CVD outcomes are not feasible.

Recent advances in biomarkers related to adipocyte health and NAFLD are of significant interest in PLWHIV. Fetuin A has been demonstrated to be associated with vascular calcification in those with obesity, NAFLD and metabolic syndrome. Adiponectin is another biomarker which is closely associated with adipocyte health and insulin resistance.

Multiparametric measures of ectopic fat (MRS, Fiborscan), cardiac structure and function (CMR), adipocyte health biomarkers (using tissue, serum and plasma) in association with CVD risk have not been studied in the same setting. We have designed this detailed cross-sectional analysis comparing PLWHIV to risk-matched general groups to inform on the role of ectopic fat in CVD in PLWHIV. This is of critical importance to gain mechanistic insight into the excess CVD risk seen in PLWHIV whilst also providing potential therapeutic targets for emerging drugs.

The increasing morbidity and mortality that CVD represents in this ageing group is of pressing concern. It represents an emerging health economic challenge for already stretched Western healthcare systems. Understanding HIV-specific mechanistic drivers of the excess CVD risk and potential therapeutic targets is therefore highly desirable. Our data and others suggest an important role for altered energy metabolism causing increased ectopic fat deposition. The development and realisation of specific therapeutics, that reduce ectopic and visceral fat, is of great interest for risk reduction strategies specifically for PLWHIV. Further understanding of the link between ectopic fat and CVD is required prior to embarking on randomised control trials for these agents. We have designed a comprehensive cross-sectional analysis investigating the associations of ectopic and visceral fat (multiple measures), intramyocardial lipid (cardiac MR spectroscopy), cardiac structure and function (CMR), biomarkers specific to energy metabolism (serum/plasma biomarkers), adipocyte health (tissue) with incident CVD (cardiovascular CT) in HIV-positive and HIV-negative / general population individuals.

The use of multiple measures of ectopic fat, including biomarkers for adipocyte health in serum and tissue, with incident CVD has not been done before. We anticipate that the data generated from this study will inform power calculations for future randomised control studies investigating the use of therapeutics on ectopic fat reduction in PLWHIV.

We have designed a cross sectional study to assess the relationship between EAT volume and CVD risk in PLWHIV and general populations. Participants will be recruited from the regional HIV service hosted by LUHFT. HIV-negative / general population participants will be recruited from those undergoing CT Coronary Angiography.

The study will involve 50 HIV-positive subjects and 50 general subjects. HIV-positive subjects will be recruited from follow up clinics and will have stable HIV disease (VL<40 copies/ml) and CD4 counts >200cells/mm3 for a minimum of 1 year. All subjects will be required to read the patient information leaflet and sign the consent form before enrolment to the study. Participants will be stratified into low (n=10), moderate (n=20) and high (n=20) risk according to traditional scoring methods. We will also include within these numbers 20 subjects with documented weight gain on INSTI regimes.

ELIGIBILITY:
Inclusion Criteria:

* • >40 years

  * HIV-positive
  * Stable ART for >6 months with two VL <40 copies/ml based on local testing protocols
  * CD4 count >200cells/mm3 for >2 years from recruitment Inclusion Criteria (all)
  * Understand the study procedures, able to comply with study procedures and voluntarily agree to participate by giving informed written consent

Exclusion Criteria:

* Subjects unable to comply with the study protocol
* History of severe renal impairment (eGFR <30ml/min)
* History of severe hepatic impairment (Child Pugh Score >9)
* Active hepatitis B or hepatitis C
* Any active illness, which in the opinion of the investigator precludes participation in the study.
* History of cancer
* Active illicit intravenous drug use
* Investigators may decide the subject cannot proceed if there are any relevant other abnormal results in screening assessments
* History or current GLP-1 agonist use
* For female subjects: pregnancy or breast feeding at screening.
* Subjects currently taking: Atypical antipsychotics, omega 3 supplements, Telmisartan/Irbesartan, Thiazolidinediones or regular NSAID use.
* Familial hypercholesterolaemia

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 participants from HIV clinic 50 participants from general population (patients undergoing CT Coronary Angiography for investigation of chest pain)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Epicardial adipose tissue volume | Through study completion, an average of 1 year
  Epicardial adipose tissue volume measured by cardiac MRI (mm3). Measurment of fat around the heart

SECONDARY OUTCOMES:
Intramyocardial triglyceride | through study completion, an average of 1 year
  MR spectroscopy. MEasurement of concentration of intramyocardial lipid content
Liver fat percentage | through study completion, an average of 1 year
  As described my MRI spectroscopy protocol. Measurement of fat content of liver cells
LV ejection fraction | through study completion, an average of 1 year
  As defined on cardiac MRI (%). Cardiac performance
Global native myocardial T1 times | through study completion, an average of 1 year
  As defined on cardiac MRI (ms). Measure of myocardial fibrosis
Lipids | through study completion, an average of 1 year
  total cholesterol (mmol/L), high density cholesterol (mmol/L), low density cholesterol (mmol/L), triglyceride (mmol/L)
LV strain on MRI | through study completion, an average of 1 year
  As defined on cardiac MRI (%). Parameter for myocardial performance
HBA1c | through study completion, an average of 1 year
  Biomarkers for insulin metabolic health(mmol/L)
Adiponectin | through study completion, an average of 1 year
  Biomarkers for insulin metabolic health (ug/ml),
Insulin | through study completion, an average of 1 year
  Biomarkers for insulin metabolic health(uU/ml)
Health status | through study completion, an average of 1 year
  Follow up will be remotely completed to record new diagnoses from electronic records for 5years.
CAP score | through study completion, an average of 1 year
  Fibroscan (dB/m). Measurement of liver fibrosis / fat

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Liverpool University Hospital, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
We will evaluate upon reasonable request to share study data (anonymised)

REFERENCES:
- [Background] Trepanowski JF, Mey J, Varady KA. Fetuin-A: a novel link between obesity and related complications. Int J Obes (Lond). 2015 May;39(5):734-41. doi: 10.1038/ijo.2014.203. Epub 2014 Dec 3. PMID 25468829
- [Background] Toribio M, Neilan TG, Awadalla M, Stone LA, Rokicki A, Rivard C, Mulligan CP, Cagliero D, Fourman LT, Stanley TL, Ho JE, Triant VA, Burdo TH, Nelson MD, Szczepaniak LS, Zanni MV. Intramyocardial Triglycerides Among Women With vs Without HIV: Hormonal Correlates and Functional Consequences. J Clin Endocrinol Metab. 2019 Dec 1;104(12):6090-6100. doi: 10.1210/jc.2019-01096. PMID 31393564
- [Background] Thirunavukarasu S, Jex N, Chowdhary A, Hassan IU, Straw S, Craven TP, Gorecka M, Broadbent D, Swoboda P, Witte KK, Cubbon RM, Xue H, Kellman P, Greenwood JP, Plein S, Levelt E. Empagliflozin Treatment Is Associated With Improvements in Cardiac Energetics and Function and Reductions in Myocardial Cellular Volume in Patients With Type 2 Diabetes. Diabetes. 2021 Dec;70(12):2810-2822. doi: 10.2337/db21-0270. Epub 2021 Oct 5. PMID 34610982
- [Background] Soares C, Kwok M, Boucher KA, Haji M, Echouffo-Tcheugui JB, Longenecker CT, Bloomfield GS, Ross D, Jutkowtiz E, Sullivan JL, Rudolph JL, Wu WC, Erqou S. Performance of Cardiovascular Risk Prediction Models Among People Living With HIV: A Systematic Review and Meta-analysis. JAMA Cardiol. 2023 Feb 1;8(2):139-149. doi: 10.1001/jamacardio.2022.4873. PMID 36576812
- [Background] Smit M, Brinkman K, Geerlings S, Smit C, Thyagarajan K, Sighem Av, de Wolf F, Hallett TB; ATHENA observational cohort. Future challenges for clinical care of an ageing population infected with HIV: a modelling study. Lancet Infect Dis. 2015 Jul;15(7):810-8. doi: 10.1016/S1473-3099(15)00056-0. Epub 2015 Jun 9. PMID 26070969
- [Background] Shah ASV, Stelzle D, Lee KK, Beck EJ, Alam S, Clifford S, Longenecker CT, Strachan F, Bagchi S, Whiteley W, Rajagopalan S, Kottilil S, Nair H, Newby DE, McAllister DA, Mills NL. Global Burden of Atherosclerotic Cardiovascular Disease in People Living With HIV: Systematic Review and Meta-Analysis. Circulation. 2018 Sep 11;138(11):1100-1112. doi: 10.1161/CIRCULATIONAHA.117.033369. PMID 29967196
- [Background] Scheuermann-Freestone M, Madsen PL, Manners D, Blamire AM, Buckingham RE, Styles P, Radda GK, Neubauer S, Clarke K. Abnormal cardiac and skeletal muscle energy metabolism in patients with type 2 diabetes. Circulation. 2003 Jun 24;107(24):3040-6. doi: 10.1161/01.CIR.0000072789.89096.10. Epub 2003 Jun 16. PMID 12810608
- [Background] Williams MC, Golay SK, Hunter A, Weir-McCall JR, Mlynska L, Dweck MR, Uren NG, Reid JH, Lewis SC, Berry C, van Beek EJ, Roditi G, Newby DE, Mirsadraee S. Observer variability in the assessment of CT coronary angiography and coronary artery calcium score: substudy of the Scottish COmputed Tomography of the HEART (SCOT-HEART) trial. Open Heart. 2015 May 19;2(1):e000234. doi: 10.1136/openhrt-2014-000234. eCollection 2015. PMID 26019881
- [Background] Mancio J, Azevedo D, Saraiva F, Azevedo AI, Pires-Morais G, Leite-Moreira A, Falcao-Pires I, Lunet N, Bettencourt N. Epicardial adipose tissue volume assessed by computed tomography and coronary artery disease: a systematic review and meta-analysis. Eur Heart J Cardiovasc Imaging. 2018 May 1;19(5):490-497. doi: 10.1093/ehjci/jex314. PMID 29236951
- [Background] Levelt E, Rodgers CT, Clarke WT, Mahmod M, Ariga R, Francis JM, Liu A, Wijesurendra RS, Dass S, Sabharwal N, Robson MD, Holloway CJ, Rider OJ, Clarke K, Karamitsos TD, Neubauer S. Cardiac energetics, oxygenation, and perfusion during increased workload in patients with type 2 diabetes mellitus. Eur Heart J. 2016 Dec 7;37(46):3461-3469. doi: 10.1093/eurheartj/ehv442. Epub 2015 Sep 20. PMID 26392437
- [Background] Le Jemtel TH, Samson R, Ayinapudi K, Singh T, Oparil S. Epicardial Adipose Tissue and Cardiovascular Disease. Curr Hypertens Rep. 2019 Apr 5;21(5):36. doi: 10.1007/s11906-019-0939-6. PMID 30953236
- [Background] Hulten E, Villines TC, Cheezum MK, Berman DS, Dunning A, Achenbach S, Al-Mallah M, Budoff MJ, Cademartiri F, Callister TQ, Chang HJ, Cheng VY, Chinnaiyan K, Chow BJ, Cury RC, Delago A, Feuchtner G, Hadamitzky M, Hausleiter J, Kaufmann PA, Kim YJ, Leipsic J, Lin FY, Maffei E, Plank F, Raff GL, Shaw LJ, Min JK; CONFIRM Investigators. Calcium score, coronary artery disease extent and severity, and clinical outcomes among low Framingham risk patients with low vs high lifetime risk: results from the CONFIRM registry. J Nucl Cardiol. 2014 Feb;21(1):29-37; quiz 38-9. doi: 10.1007/s12350-013-9819-7. Epub 2014 Jan 3. PMID 24385134
- [Background] Hulgan T, Ramsey BS, Koethe JR, Samuels DC, Gerschenson M, Libutti DE, Sax PE, Daar ES, McComsey GA, Brown TT. Relationships Between Adipose Mitochondrial Function, Serum Adiponectin, and Insulin Resistance in Persons With HIV After 96 Weeks of Antiretroviral Therapy. J Acquir Immune Defic Syndr. 2019 Mar 1;80(3):358-366. doi: 10.1097/QAI.0000000000001926. PMID 30531304
- [Background] Holloway CJ, Ntusi N, Suttie J, Mahmod M, Wainwright E, Clutton G, Hancock G, Beak P, Tajar A, Piechnik SK, Schneider JE, Angus B, Clarke K, Dorrell L, Neubauer S. Comprehensive cardiac magnetic resonance imaging and spectroscopy reveal a high burden of myocardial disease in HIV patients. Circulation. 2013 Aug 20;128(8):814-22. doi: 10.1161/CIRCULATIONAHA.113.001719. Epub 2013 Jul 1. PMID 23817574
- [Background] Heseltine T, Murray S, Ortega-Martorell S, Olier I, Lip GYH, Khoo S. Associations of Hepatosteatosis With Cardiovascular Disease in HIV-Positive and HIV-Negative Patients: The Liverpool HIV-Heart Project. J Acquir Immune Defic Syndr. 2021 Aug 15;87(5):1221-1227. doi: 10.1097/QAI.0000000000002721. PMID 33990492
- [Background] Heseltine T, Hughes E, Mattew J, Murray S, Ortega-Martorell S, Olier I, Dey D, Lip GYH, Khoo S. The association of epicardial adipose tissue volume and density with coronary calcium in HIV-positive and HIV-negative patients. J Infect. 2023 Apr;86(4):376-384. doi: 10.1016/j.jinf.2023.02.020. Epub 2023 Feb 16. PMID 36801347
- [Background] Goeller M, Achenbach S, Marwan M, Doris MK, Cadet S, Commandeur F, Chen X, Slomka PJ, Gransar H, Cao JJ, Wong ND, Albrecht MH, Rozanski A, Tamarappoo BK, Berman DS, Dey D. Epicardial adipose tissue density and volume are related to subclinical atherosclerosis, inflammation and major adverse cardiac events in asymptomatic subjects. J Cardiovasc Comput Tomogr. 2018 Jan-Feb;12(1):67-73. doi: 10.1016/j.jcct.2017.11.007. Epub 2017 Nov 24. PMID 29233634
- [Background] Garrabou G, Lopez S, Moren C, Martinez E, Fontdevila J, Cardellach F, Gatell JM, Miro O. Mitochondrial damage in adipose tissue of untreated HIV-infected patients. AIDS. 2011 Jan 14;25(2):165-70. doi: 10.1097/QAD.0b013e3283423219. PMID 21150553
- [Background] Eisenberg E, McElhinney PA, Commandeur F, Chen X, Cadet S, Goeller M, Razipour A, Gransar H, Cantu S, Miller RJH, Slomka PJ, Wong ND, Rozanski A, Achenbach S, Tamarappoo BK, Berman DS, Dey D. Deep Learning-Based Quantification of Epicardial Adipose Tissue Volume and Attenuation Predicts Major Adverse Cardiovascular Events in Asymptomatic Subjects. Circ Cardiovasc Imaging. 2020 Feb;13(2):e009829. doi: 10.1161/CIRCIMAGING.119.009829. Epub 2020 Feb 17. PMID 32063057
- [Background] Cho I, Al'Aref SJ, Berger A, O Hartaigh B, Gransar H, Valenti V, Lin FY, Achenbach S, Berman DS, Budoff MJ, Callister TQ, Al-Mallah MH, Cademartiri F, Chinnaiyan K, Chow BJW, DeLago A, Villines TC, Hadamitzky M, Hausleiter J, Leipsic J, Shaw LJ, Kaufmann PA, Feuchtner G, Kim YJ, Maffei E, Raff G, Pontone G, Andreini D, Marques H, Rubinshtein R, Chang HJ, Min JK. Prognostic value of coronary computed tomographic angiography findings in asymptomatic individuals: a 6-year follow-up from the prospective multicentre international CONFIRM study. Eur Heart J. 2018 Mar 14;39(11):934-941. doi: 10.1093/eurheartj/ehx774. PMID 29365193
- [Background] Cheney L, Hou JC, Morrison S, Pessin J, Steigbigel RT. Nef inhibits glucose uptake in adipocytes and contributes to insulin resistance in human immunodeficiency virus type I infection. J Infect Dis. 2011 Jun 15;203(12):1824-31. doi: 10.1093/infdis/jir170. PMID 21606541
- [Background] Agarwal N, Iyer D, Patel SG, Sekhar RV, Phillips TM, Schubert U, Oplt T, Buras ED, Samson SL, Couturier J, Lewis DE, Rodriguez-Barradas MC, Jahoor F, Kino T, Kopp JB, Balasubramanyam A. HIV-1 Vpr induces adipose dysfunction in vivo through reciprocal effects on PPAR/GR co-regulation. Sci Transl Med. 2013 Nov 27;5(213):213ra164. doi: 10.1126/scitranslmed.3007148. PMID 24285483